CLINICAL TRIAL: NCT05034549
Title: Efficacy and Safety of Home Non-invasive Ventilation Based on Polysomnography in Chronic Stable Heart Failure
Brief Title: Noninvasive Ventilation for Chronic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Pan-Pan Hao, MD, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Qilu-CHF
Record Dates: First submitted 2020-11-08; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Chronic Stable Heart Failure
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Noninvasive ventilation (Experimental)
  Interventions: Device: Noninvasive ventilation

INTERVENTIONS:
Device: Noninvasive ventilation — The non-invasive ventilator at home (≥5h/ night)
  Arms: Noninvasive ventilation

SUMMARY:
The effects of home noninvasive ventilation on renin-angiotensin system (RAS), kallikrein-kinin system (KKS) and cardiac remodeling in patients with chronic stable heart failure have not been reported. This project aims to clarify the efficacy and safety of home non-invasive ventilation in patients with chronic heart failure complicated with sleep-disordered breathing. First, patients with chronic stable heart failure were selected and monitored by polysomnography. Patients with sleep apnea hypopnea syndrome (SAHS, AHI≥15) were randomly divided into two groups: the treatment group was treated with non-invasive ventilator at home (≥5h/ night); The control group was only given routine treatment. After 6 months of follow-up, the effects of sleep disordered breathing and noninvasive ventilation on RAS, KKS, cardiac remodeling and function and cardiovascular adverse events in patients with chronic heart failure were evaluated. The results are helpful to further reveal the role of sleep disordered breathing in the occurrence and development of chronic heart failure, and provide a new diagnosis and treatment strategy for chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* 1) The history of chronic stable heart failure exceeds 3 months; 2) 18~75 years old; 3) NYHA cardiac function classified as grade II~IV; 4) LVEF≤40%； 5) NT-proBNP≥450pg/ml； 6) All subjects or their guardians must sign the subject consent before entering the trial.

Exclusion Criteria:

* 1) Patients with the following diseases: valvular heart disease; congenital heart disease; obstruction of left ventricular outflow tract; severe decompensated heart failure; acute coronary syndrome; active myocarditis or pericardial disease; end-stage liver and kidney diseases; malignant tumor; 2) Patients with poor sound transmission windows are examined by transthoracic ultrasound.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Cardiac remodeling | 6 months
  The difference of left ventricular end diastolic volume (LVEDV) compared with baseline

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Qilu Hospital, Shandong University, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong
  - Jinan Central Hospital Affiliated to Shandong First Medical University, Jinan

IPD SHARING:
Plan to Share IPD: No